CLINICAL TRIAL: NCT07174141
Title: Innovative Biomarkers of Cardiovascular Complications Associated With Second-generation Bruton Tyrosine Kinase Inhibitor Treatments: a Single-center Cohort Study
Acronym: CACIS II
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ROBERT_AOI_2022
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Treatment With Second-generation Bruton's Tyrosine Kinase Inhibitors (Acalabrutinib, Zanubrutinib)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients: Patients eligible for treatment with second-generation Bruton's tyrosine kinase inhibitors in hematology (acalabrutinib, zanubrutinib)
  Interventions: Other: Ophthalmological examination; Biological: Blood sample

INTERVENTIONS:
Other: Ophthalmological examination — at inclusion, at 3 months and 6 months; OCT-A retina
Biological: Blood sample — Collection of a 2 mL blood sample at inclusion

SUMMARY:
Second-generation Bruton's tyrosine kinase inhibitors (BTKIs) (zanubrutinib, acalabrutinib) are recently discovered oral targeted therapies used to treat hematological disorders such as chronic lymphocytic leukemia, mantle cell lymphoma, non-Hodgkin's lymphoma, and Waldenström's macroglobulinemia.

These treatments significantly increase survival rates for these diseases, but over the years, we have observed the emergence of cardiovascular adverse effects such as cardiac arrhythmia and high blood pressure, the type and frequency of which differ from those of first-generation drugs such as ibrutinib.

The frequency of these cardiovascular events remains poorly understood, as do the risk factors for developing these complications.

The aim of this study is to determine the exact incidence of cardiac arrhythmia and high blood pressure in patients receiving second-generation IBTK and to identify risk factors that can predict these complications through close, specialized monitoring.

Ultimately, this will make it possible to better target patients at highest risk of developing cardiovascular complications and offer them appropriate follow-up care.

This is a single-center, prospective, observational study conducted at the Dijon Bourgogne University Hospital.

The required number of subjects is 100 patients. The total follow-up period for each patient is one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment with second-generation Bruton's tyrosine kinase inhibitors in hematology (acalabrutinib, zanubrutinib)
* Patients aged 18 years and older
* Patients who have given their free and informed written consent to participate in this study after receiving information (or the patient's representative if the patient is unable to express consent themselves).
* Patients with a life expectancy estimated by the hematologist in charge of the patient to be greater than one year

Exclusion Criteria:

* Persons not affiliated with or not covered by a social security system
* Patients subject to legal protection measures (guardianship, trusteeship)
* Patients subject to judicial protection measures
* Pregnant women, women in labor, or breastfeeding women
* Prior treatment with Bruton's tyrosine kinase inhibitors (ibrutinib, acalabrutinib, zanubrutinib)
* Follow-up planned at another center
* History of atrial fibrillation
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for treatment with second-generation Bruton's tyrosine kinase inhibitors in hematology (acalabrutinib, zanubrutinib)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a diagnosis of new-onset high blood pressure or worsening of pre-existing hypertension | 12 months after initiation of treatment with second-generation Bruton's tyrosine kinase inhibitors in hematology

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France